CLINICAL TRIAL: NCT03567512
Title: Reducing Second-hand Smoke Exposure Among Young Children in Rural China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Taizhou Municipal Center for Disease Control and Prevention (Unknown); Fudan University (Other)
Responsible Party: Principal Investigator, Abu Abdullah, Professor, Duke Kunshan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 71673125
Record Dates: First submitted 2018-06-06; First posted 2018-06-25 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Second Hand Tobacco Smoke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Intervention administered to this group will focus on Quit Smoking of parental and household smokers and Reduction of Secondhand Smoke Exposure among the Children.
  Interventions: Behavioral: Smoking hygiene intervention
- Control group (Placebo Comparator): The placebo intervention will be administered in this group.
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Smoking hygiene intervention — The Smoking Hygiene Intervention(SHI) will be delivered in six different individualized counseling sessions (two in-person and four telephone counseling): the initial in-person counseling (30-45 minutes), 1 week telephone counseling (~20 minutes), 2 week telephone counseling (~20 minutes), 1 month in-person counseling (15-30 minutes), 2 month telephone counseling (~20 minutes), and 4 month telephone counseling (~20 minutes). The intervention, SHI, will address SHS exposure of children and parental quitting. It will include behavioral counseling to address health hazards of SHS for children, advice to quit smoking and to adopt a no smoking policy around children and self-help materials (related to second-hand smoking and quitting smoking).
  Arms: Intervention group
Behavioral: Placebo intervention — The placebo intervention will include developmental perspective of the child at different stages of their life, advice on educational and emotional perspective of the child, discussion on the nutritional issues of the child, and self-help materials describing the child development issues.
  Subjects randomized to control group will receive a placebo intervention on child development issues delivered at six different individualized counseling sessions (two in-person and four telephone counseling): the initial in-person counseling (30-45 minutes), 1 week telephone counseling (~20 minutes), 2 week telephone counseling (~20 minutes), 1 month in-person counseling (15-30 minutes), 2 month telephone counseling (~20 minutes), and 4 month telephone counseling (~20 minutes).
  Arms: Control group

SUMMARY:
Second-hand smoking (SHS) is a health hazard to infants and children, in whom it is associated with lower respiratory tract infections, wheezing, cough, middle ear infections and sudden infant death syndrome. The high prevalence of smoking in adults in China, 52.9% among men, 2.4% among women, results in many children being exposed to SHS at home. Data on the effectiveness of evidence-based smoking hygiene intervention to reduce SHS exposure among young children (e.g., aged 5 or below) is lacking in China. Children in the rural setting are more exposed to SHS due to the lack of tobacco control policy initiative in the rural setting and the high prevalence of smoking among the rural public. In the proposed project we aim to examine the effectiveness of a protection motivation theory-based smoking hygiene intervention (SHI), delivered by community health worker (CHW) in 6 different contacts, to reduce SHS exposure among young children in two rural areas of China: Taizhou city (Zhejiang Province) and Dali city (Yunnan province). The results of this study will provide clinical evidence for the development of CHW-delivered interventions designed to reduce exposure to SHS and related morbidity and mortality among children in rural China. The successful results could also be used to draft guidelines for health promotion interventions, which could be implemented as a policy for all primary health care settings in rural China and other developing countries.

DETAILED DESCRIPTION:
Second-hand smoking (SHS) is a health hazard to infants and children, in whom it is associated with lower respiratory tract infections, wheezing, cough, middle ear infections and sudden infant death syndrome. With a population of 1.2 billion, China is the world's largest producer and consumer of tobacco, with over 350 million smokers. The high prevalence of current smoking among men (60.2%) and women (6.9%) in China, reflect the fact that a large number of young children are exposed to SHS at home. The high exposure to SHS increases children's risk of tobacco-induced morbidity and mortality. Children in the rural setting even are more exposed to SHS due to the lack of tobacco control policy initiative in the rural setting and the high prevalence of smoking among the rural public.

While evidence-based intervention to reduce children's exposure to SHS was proven effective in the United States, data on the effectiveness of evidence-based interventions to reduce SHS exposure among young children (e.g., under age 5) is lacking in rural China.

China's unique public health history and homogeneity of the population provide an unprecedented opportunity to examine the effects of an exposure reduction intervention (we will call this as "smoking hygiene intervention, SHI") among children. Community health workers (CHWs), who play an important role in delivering other health interventions (i.e. vitamin supplementation and treatment for acute respiratory infection), offer a resource for delivery of SHI intervention in the community level.

To address this growing problem and to develop local evidence base, the proposed study will examine the effectiveness of a protection motivation theory (PMT) -based SHI, delivered by community health worker (CHW) in 6 different contacts, to reduce SHS exposure among young children and promote parental quitting in two rural setting of Zhejiang and Shanxi provinces. The results of this study will provide clinical evidence for the development of CHW-delivered interventions designed to reduce exposure to SHS and related morbidity and mortality among children in rural China. The successful results could also be used to draft guidelines for health promotion interventions, which could be implemented as a policy for all primary health care settings in rural China and other developing countries.

The study population will consist of the smoker household members of young children aged 5 years or below in the selected community. Families with at least one smoker in the household (mother, father or other household members) will be invited to participate in the intervention study. Investigators will recruit a total of 400 smoker household members; 200 from rural Zhejiang province and 200 from rural Yunnan province (Dali district).

Methodology:

The study will be divided into two parts. The first is a baseline assessment study. The second is a randomized controlled trial (RCT) of households in the targeted community.

1. Baseline assessment:

   The aim of the baseline assessment is to obtain baseline data on second-hand tobacco exposure among young children, the health status of children and smoking status of household members, and to screen and offer an invitation to participate in the study. A structured questionnaire, after pilot testing, will be used for data collection. A brief screening form to assess eligibility for intervention study will also be completed during the baseline assessment. All the collected screening forms, both eligible and not eligible, will be kept in the research office and will follow the institutional data storage and safety procedures.

   Investigators will recruit four interviewers to work on this project. Interviewers will collect baseline data and the follow-up data at 2 months and 6 months. Interviewers will forward all of their collected data on a weekly basis to a central data supervisor based at participating collaborating institutions. Interviewers will also do the followings: measure carbon monoxide (CO) level in exhaled air of those smokers who reportedly quitted smoking (at 2-and 6-months), and collect child's urine samples for cotinine measures. Criteria for the interviewer will be (1) at least higher secondary school graduate, (2) ability to speak and read Mandarin Chinese fluently, (3) ability to speak local (Taizhou or Dali) dialect and (4) familiarity with the populations in which they will be working.

   Training of interviewer: Interviewers will receive training on: (a) Research ethics to ensure that they follow the guidelines of the US NIH standard and Duke Kunshan guidelines to collect data, (b) data collection methods, (c) measuring carbon monoxide level in exhaled air, (d) collection of urine samples, and (e) storage of urine samples in cool box. The intensive 1-day training will be provided by the investigators and will be conducted in Chinese.

   The training will provide them with the necessary communication and interview skills so that they can conduct successful interviews and collect useful data. During the training, the interviewers will be taken through the questionnaire question by question, explaining them thoroughly and the information required. They will also perform mock testing to measure CO in exhaled air and collection and storage of urine samples. Training methods that will be used will include, discussions, practice and role play.
2. Randomized controlled trial (RCT).

To collect preliminary data regarding the intervention's effectiveness we will conduct an RCT. After confirming the eligibility criteria and informed consent, the household members will be randomly allocated to either the intervention group or the control group. Randomization will be done by opening a serially labeled opaque and sealed envelope with a card indicating the randomly allocated group (i.e. A= Intervention group, B= Control group). The trial will begin as soon as the baseline assessment has been completed and the relevant institutes have given ethical approval.

Follow-up assessment: Follow-up will be carried out at 2 months and 6 months after initial contact for both the intervention and control group. The 2-month and 6-month follow up data will be collected by interviewers who will be blinded to the study conditions of the households. Each follow-up assessment will last about 30 minutes. At 2 month follow-up, the household smoking practices, health-related information of children and the smoking status of all subjects will be assessed by interviewers through face-to-face interview using the standard questionnaire. At 6 month follow-up, all subjects will be contacted by interviewers for final assessment through a face-to-face interview. Their household smoking practices, smoking and quitting related information and health-related information of child will be collected using the standard questionnaire.

Community Health Worker (CHW): Intervention will be provided by CHWs who have been working in the relevant community centers for at least 3 months. CHWs will be literate (at least a higher secondary school degree), have participated in community work or clinical work for children, and be fluent in both the local dialect and Mandarin Chinese. After training, they must be competent in counseling parents of young children or other household members on SHI. CHWs must be available and willing to visit households to deliver interventions at subjects' homes or other convenient facilities within the community.

Training of CHW: CHWs will be trained on SHI. Guidelines will be developed detailing the SHI. The intensive 2-day training (8 hours each) will be provided by the investigators and will be conducted in Chinese. The curriculum for the training will include the following key components: (i) health consequences of smoking and SHS. It will emphasize the acute health effects of secondhand smoke on children, especially regarding the development of asthma, exacerbation of existing asthma, middle ear infections, upper respiratory infections, and perhaps the relationship between secondhand smoke exposure and sudden infant death syndrome (SIDS). These would be key components of the training so that the workers truly understand the devastating impact that secondhand smoke can have on the health of these children, and so that when intervening with parents, they can emphasize these health effects accurately, (ii) benefits of reducing children's exposure to SHS. It will discuss both health and economic benefits and use real-life examples to illustrate the fact; (iii) understanding child development issues in different stages of childhood; iv) basic counseling skills; v) motivational enhancement strategies; (vi) assessment of smoking status using CO monitor, and vi) study procedures.

Performance assessment of CHW: The assessment of the performance of the CHWs is very crucial to the success of the study. This will allow us to find out whether the CHWs still possess the skills obtained during the training and are being used. The assessment of their performance will be done through the following methods in every two months during the 6 months of the intervention period. The first will be done through the random examination of the action plan (i.e. summary note) being kept by the CHW for each subject. From the action plan, supervisors can indicate whether CHWs are providing intervention based on the protocol and whether the appropriate measures were taken based on the problems noted in the action plan. The supervisor will also assess the performance of CHWs by observing them while counseling household members. The supervisor will accompany CHW and observe at least 2 counseling sessions. The report of these assessments will be compiled by the supervisor and reviewed by investigators to determine whether there is need of refresher course for the CHWs.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above) household member has smoked one or more cigarettes daily for the past 30 days as self-reported;
* household smoker smokes a total of at least 10 cigarettes per week at home in the presence of the child, as self-reported;
* smoker household member and the child are living together in the same household and will live together during the entire period of the study;
* residents of the study community, (v) able to communicate in Mandarin Chinese;
* has signed an informed consent form or given verbal consent (for those who cannot read and write);
* willing to give urine sample of the child for biochemical measures.

Exclusion Criteria:

* household members do not smoke at home;
* smoker member does not live in the same household as the child;
* non-local community resident, and (iv) not able to communicate in Mandarin Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in the smoking hygiene practices | At 6 month after intervention
  Changes in smoking hygiene practices within the household as reported by the subjects (ie, adoption of complete smoking restriction at home (yes/no), and change in the exposure of SHS to child from household members inside the home as measured by exposure to mean number of cigarettes per week)

SECONDARY OUTCOMES:
Change of respiratory illness incidence | At 6 month after intervention
  Change of, from baseline to at 6-months, respiratory illness incidence among children as reported by key household member
Self-reported parental quit smoking | At 6 months after intervention
  Not smoking any cigarette in the past 7 days at 6-moths follow up, as reported by the participants.
Change of urine cotinine concentration | At 2 and 6 momths
  Change of mean urine cotinine concentration from baseline to at 2 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abu Abdullah, PhD, Study Chair — Duke Kunshan University
Locations (1):
- Taizhou Municipal center for disease control and prevention, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiFranza JR, Lew RA. Morbidity and mortality in children associated with the use of tobacco products by other people. Pediatrics. 1996 Apr;97(4):560-8. PMID 8632946
- [Background] Mannino DM, Siegel M, Husten C, Rose D, Etzel R. Environmental tobacco smoke exposure and health effects in children: results from the 1991 National Health Interview Survey. Tob Control. 1996 Spring;5(1):13-8. doi: 10.1136/tc.5.1.13. PMID 8795853
- [Background] American Academy of Pediatrics. Involuntary smoking--a hazard to children. Committee on Environmental Hazards. Pediatrics. 1986 May;77(5):755-7. No abstract available. PMID 3703641
- [Background] Yao T, Sung HY, Mao Z, Hu TW, Max W. Secondhand smoke exposure at home in rural China. Cancer Causes Control. 2012 Mar;23 Suppl 1(0 1):109-15. doi: 10.1007/s10552-012-9900-6. Epub 2012 Feb 12. PMID 22327886